CLINICAL TRIAL: NCT02295969
Title: An Observational Study of ORALAIR® (Grass Pollen Allergen Extract From: Cocksfoot, Sweet Vernal, Rye Grass, Meadow Grass, Timothy) Tablet for Sublingual Use in Children 5 to 9 Years of Age With Grass-pollen-induced Allergic Rhinitis With or Without Conjunctivitis
Brief Title: Observational Study of Oralair® in Children 5-9 Years With Grass-pollen-induced Allergic Rhinitis With/Without Conjunctivitis
Status: Completed | Type: Observational
Sponsor: Stallergenes Greer (Industry)
Collaborators: Venn Life Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: SL74.14
Record Dates: First submitted 2014-11-18; First posted 2014-11-20 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Allergy
Keywords: Rhinitis; Conjunctivitis; Grass pollen; Sublingual tablet; Allergen immunotherapy; Safety
MeSH Terms: conditions — Hypersensitivity; Rhinitis; Conjunctivitis | interventions — Sweet Vernal, orchard, Perennial Rye, Timothy and Kentucky Blue Grass Mixed Pollens Allergen Extract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Oralair — Observational study, Oralair is used as prescribed by the prescriber phycisian.

SUMMARY:
Safety and tolerability of ORALAIR in children 5 to 9 years of age during the first 30 days of treatment.

DETAILED DESCRIPTION:
The purpose of this study is to further describe the safety and tolerability of ORALAIR tablets in children 5 to 9 years of age with grass-pollen-induced allergic rhinitis with or without conjunctivitis.

Patients are followed for safety and tolerability during the first 30 treatment days.

ELIGIBILITY:
Inclusion Criteria:

Allergen immunotherapy naive male or female outpatients aged 5 to 9 years (inclusive) prescribed ORALAIR.

Exclusion Criteria:

Patients already participating in a clinical trial.

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Outpatients, children 5 to 9 years of age prescribed ORALAIR for the treatment of grass-pollen-induced allergic rhinitis with or without conjunctivitis.
Sampling Method: Non-Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2014-12; Primary Completion 2017-07-03 (Actual); Study Completion 2017-07-03 (Actual)

PRIMARY OUTCOMES:
All adverse events that started on or after the day the first dose of Oralair | During 30 days after the date of the first dose

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum Augsburg, Klinik für Kinder und Jugendliche, Augsburg, Bavaria, Germany

REFERENCES:
- [Derived] Gerstlauer M, Szepfalusi Z, Golden D, Geng B, de Blic J. Real-life safety of 5-grass pollen tablet in 5-to-9-year-old children with allergic rhinoconjunctivitis. Ann Allergy Asthma Immunol. 2019 Jul;123(1):70-80. doi: 10.1016/j.anai.2019.04.011. Epub 2019 Apr 19. PMID 31009701